CLINICAL TRIAL: NCT06908304
Title: A Multicenter, Open-label, Randomized Phase 3 Study of THIO Sequenced With Cemiplimab (LIBTAYO®) vs Investigator's Choice of Chemotherapy as Third-line Treatment in Advanced/Metastatic NSCLC
Brief Title: A Phase III Study With THIO + Cemiplimab vs Chemotherapy as 3rd Line Treatment in Advanced/Metastatic NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maia Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THIO-104; 2024-520164-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small -Cell Lung
Keywords: squamous cell carcinoma; Adenocarcinoma; Non-Small Cell Lung Carcinoma; Non-Small Cell Lung Cancer; Large Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Large Cell | interventions — alpha-2'-deoxythioguanosine; cemiplimab; Docetaxel; Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- THIO + Cemiplimab Arm (Experimental): THIO 60mg, 30-min IV infusions, Days 1-3 (180 mg/Cycle) Cemplimab 350 mg, 30-min IV infusion, Day 5
  3-Week Cycle
  Interventions: Drug: 6-Thio-2'-Deoxyguanosine; Drug: Cemiplimab
- Investigator's choice of single-agent chemotherapy (vinorelbine, gemcitabine, or docetaxel) (Active Comparator): Chemotherapy Agent [1] Dosing Regimen No. of Subjects (Planned) Option 1: Vinorelbine 30 mg/m2 IV on D1, D8, and D15 Q3W ~150 [3] Option 2: Gemcitabine 1250 mg/m2 IV on D1 and D8 Q3W Option 3: Docetaxel 75 mg/m2 IV on D1 Q3W [2]
  Abbreviations: D = day (within a 21-day cycle); IV= intravenous; Q3W=every 3 weeks (21-day cycles)
  1. Standard of Care (for example vinorelbine, gemcitabine, or docetaxel chemotherapy, if not previously exposed, per Investigator's Choice)
  2. Docetaxel 60-65 mg/m2 permitted based on country-specific approvals.
  3. Within the control arm, there are no limits on the number of subjects who can be treated with any of the chemotherapy agents.
  Interventions: Drug: Docetaxel; Drug: Vinorelbine; Drug: Gemcitabine alone

INTERVENTIONS:
Drug: 6-Thio-2'-Deoxyguanosine — small molecule telomere targeting agent
  Other Names: 6-thio-dG; THIO; ateganosine
  Arms: THIO + Cemiplimab Arm
Drug: Cemiplimab — programmed cell death protein 1 (PD-1) inhibitor
  Other Names: LIBTAYO®
  Arms: THIO + Cemiplimab Arm
Drug: Docetaxel — Chemotherapy drug; inhibits cell division by stabilizing microtubules. Used for breast, lung, and prostate cancers.
  Other Names: Taxotere; Docecad
  Arms: Investigator's choice of single-agent chemotherapy (vinorelbine, gemcitabine, or docetaxel)
Drug: Vinorelbine — Chemotherapy drug; disrupts microtubule formation, inhibiting cell division. Used for non-small cell lung cancer and breast cancer.
  Other Names: Navelbine; Vinorelbine tartrate
  Arms: Investigator's choice of single-agent chemotherapy (vinorelbine, gemcitabine, or docetaxel)
Drug: Gemcitabine alone — Chemotherapy drug; inhibits DNA synthesis. Used for pancreatic, lung, breast, and ovarian cancers.
  Other Names: Gemzar
  Arms: Investigator's choice of single-agent chemotherapy (vinorelbine, gemcitabine, or docetaxel)

SUMMARY:
THIO is a first-in-class small molecule telomere targeting agent, in development for the treatment of non-small cell lung cancer (NSCLC) in combination with cemiplimab (LIBTAYO®). THIO is preferentially incorporated into telomeres sequence in telomerase-positive cells leading to rapid telomere uncapping, genomic instability, and cell death.

Cemiplimab is a programmed cell death protein 1 (PD-1) inhibitor recently approved as a first-line treatment for patients with locally advanced or metastatic NSCLC with 50% or more PD-L1 expression. It is hypothesized that THIO administration prior to cemiplimab would restore tumor responses to immunotherapy in subjects who either developed resistance or relapsed after receiving first line treatment with an immune check point inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of signing the Informed Consent Form (ICF) prior to initiation of any study specific activities/procedures.

   Disease Characteristics
2. Stage 3b or 4 histologically or cytologically confirmed NSCLC. Note: Stage is determined at the time of diagnosis.
3. Two (2) prior lines of systemic treatment for advanced/metastatic disease, including an ICI (anti-PD-1/PD-L1) and a platinum-based chemotherapy (given in combination or in separate lines) for advanced/metastatic disease.

   Note: The combination of primary therapy followed by maintenance is considered as one line of therapy. Prior treatment with docetaxel is preferred (but not mandated) and is a pre-specified stratification factor.
4. Documented progression or intolerance following the most recent line of therapy.

   * Stage 4 subjects - must have progressed or relapsed after first-line treatment.
   * Stage 3b subjects - must have already failed, or be ineligible for, local, curative-intent therapy including surgery, and/or chemoradiation.

   Note: Local, curative-intent therapy including surgery, and/or chemoradiation is not considered a treatment line in the advanced setting.
5. Documented secondary resistance to the prior ICI treatment, as defined by the SITC IRTF (Kluger, 2020):

   Resistance phenotype Drug exposure requirements Best response Confirmation scan for PD requirement Confirmation scan timeframe Secondary resistance ≥ 6 months CR, PR, SD for > 6 months Yes [1] At least 4 weeks after disease progression (per RECIST V1.1) [1] Other than when tumor growth is very rapid, and subjects are deteriorating clinically.

   Abbreviations: CR=complete response; PD=progressive disease; PR=partial response; SD=stable disease
6. No prior targeted therapy for driver mutations.
7. At least one measurable target lesion that meets the definition of RECIST v1.1, with documented progression following the most recent line of therapy.
8. An archival tissue sample (formalin fixed paraffin-embedded [FFPE] tissue block or unstained slides) is required if tissue is available at baseline.

   Note: The sample does not need to be received by the central laboratory prior to Cycle 1, Day 1 (C1D1). Subjects without archival tissue available at baseline may be eligible with Medical Monitor approval.

   Diagnostic Assessments
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
10. Demonstrate adequate organ function as defined below. All screening laboratories should be performed up to 14 days before initiating IP:

    Bone marrow function:

    ○ Neutrophil count ≥ 1500/mm3, hemoglobin ≥ 9.0 g/dL, platelet count ≥ 100,000/mm3

    Liver function:
    * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN), up to ≤ 3 × ULN if due to Gilbert's syndrome
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN.

    Note: For subjects with liver metastases present at baseline, ALT and/or AST ≤ 3 × ULN is permitted.

    Renal function:

    ○ Creatinine clearance (CrCl) ≥ 60 mL/min calculated by the Cockcroft-Gault formula using actual body weight (see Table 18) or 24-hour urine collection.

    Gender and Reproductive Requirements
11. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to receiving the first administration of IP.
12. Contraception use:

In the THIO / cemiplimab arm:

* WOCBP must agree to use a highly effective birth control and refrain from oocyte donation during the study (prior to the first dose with THIO, for the duration of the treatment with THIO, and for six months after the last dose of study treatment, if conception is possible during this interval).
* Unless permanently sterile by bilateral orchidectomy, male subjects and WOCBP partners of male subjects should use a combination of the methods specified for female subjects in Appendix 4, Section 10.4 along with a male condom, from start of study treatment, for the duration of the treatment, and for six months after the last dose of study treatment. Male subjects should also refrain from sperm donation during this time.

In the single-agent chemotherapy arm: For WOCBP, male subjects and WOCBP partners of male subjects, contraception requirements should follow the relevant product's package labelling and standard of care.

Note: Contraception use by men or women in both treatment arms should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Informed Consent 13. Capable and willing to give signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. For subjects who have received prior treatment with a checkpoint inhibitor: primary resistance to prior checkpoint inhibitor, as defined by the SITC IRTF (Kluger, 2020):

   Resistance phenotype Drug exposure requirements Best response Confirmation scan for PD requirement Confirmation scan timeframe Primary resistance ≥ 6 weeks PD; SD for < 6 months Yes [1] At least 4 weeks after initial disease progression (per RECIST v1.1) [1] Other than when tumor growth is very rapid, and subjects are deteriorating clinically.

   Abbreviations: CR=complete response; PD=progressive disease; PR=partial response; SD=stable disease Note: Subjects with drug exposure > 6 weeks who achieved a partial or complete response then progressed before six months, would still be eligible.
2. Untreated or symptomatic central nervous system (CNS) metastases. Note: Subjects with treated asymptomatic brain metastasis are eligible.
3. Prior chemotherapy and/or non-biologic targeted therapy within 28 days, or biologic targeted therapy, immunotherapy, and/or radiation therapy within 42 days prior to start of study treatment.

   Note: Subjects who receive targeted radiation therapy for localized palliative care may be eligible to start study treatment earlier than 42 days with Medical Monitor agreement.
4. Prior treatment with cemiplimab.
5. Prior treatment with a targeted therapy for an epidermal growth factor receptor (EGFR) mutation.
6. Received blood, red blood cell or platelet transfusion within 14 days prior to start of study treatment.
7. Any live, attenuated, inactivated or research vaccines within 30 days prior to start of study treatment.

   Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed.
8. Prior allogeneic hematopoietic stem cell transplant or solid organ transplant.
9. Undergone major surgery within 28 days prior to start of study treatment. Medical conditions
10. Have not recovered to Grade ≤ 1 from adverse events due to prior anti-cancer treatment.
11. Ongoing immune-related / stimulated adverse events (irAEs) from other agents or required permanent discontinuation of prior ICIs due to irAEs.

    Note: Subjects with resolved irAE may be allowed to enroll following consultation with the Medical Monitor.
12. Active gastrointestinal bleeding as evidenced by either hematemesis or melena.
13. History of another concurrent malignancy other than the present condition (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of three years.
14. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to start of study treatment.

    Note: Inhaled or topical steroids, adrenal replacement doses 10 mg daily prednisone equivalents, and systemic corticosteroids to manage adverse events are permitted in the absence of active autoimmune disease.
15. Active, uncontrolled bacterial, viral or fungal infections, requiring systemic therapy within 14 days of screening.
16. Positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active hepatitis B or hepatitis C.
17. Significant cardiovascular impairment (history of New York Heart Association Functional Classification System Class III or IV) or a history of myocardial infarction or unstable angina within the past six months prior to start of study treatment.
18. QT interval corrected for heart rate (using Fridericia's correction formula; QTcF) > 480 msec at screening (based on average of triplicate electrocardiograms [ECGs] at baseline).

    Note: If the QTc is prolonged in a subject with a pacemaker or bundle branch block, the subject may be enrolled in the study if confirmed by the Medical Monitor.
19. Active autoimmune diseases or history of autoimmune diseases that may relapse, with the following exceptions:

    * Controlled Type 1 diabetes
    * Hypothyroidism (provided it is managed with hormone replacement therapy only)
    * Controlled celiac disease
    * Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia)
    * Any other disease that is not expected to recur in the absence of external triggering factors.
20. Pregnancy or lactating.
21. A serious nonmalignant disease (e.g., psychiatric, substance abuse, uncontrolled intercurrent illness, interstitial lung disease etc.) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
22. Any other condition that, in the opinion of the Investigator, would prohibit the subject from participating in the study.

    Prior / concurrent clinical study experience
23. Currently enrolled in a clinical study involving another investigational product or nonapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

    Other
24. History of allergy to excipients of THIO, cemiplimab or any of the chemotherapies under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Within 2 Years
  Overall survival as defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Objective Radiographic Response | Within 2 Years
  Objective Radiographic Response as defined as the proportion of subjects demonstrating a confirmed objective response of complete response or partial response.
Disease Control Rate | Within 2 Years
  Disease Control Rate as defined as the proportion of subjects demonstrating complete response, partial response, or stable disease after 2 treatment cycles.
Duration of Response | Within 2 Years
  Duration of Response as defined as the time from response complete response or partial response to progressive disease.
Progressive Free Survival | Within 2 Years
  Progressive Free Survival as defined as the time from randomization to the first occurrence of progressive disease or death from any cause, whichever occurs first.
Treatment Emergent Adverse events and Serious Adverse Events | Within 2 Years
  Incidence of Treatment Emergent Adverse events and Serious Adverse Events leading to discontinuation of study medication (THIO and/or cemiplimab) and/or withdrawal from the study.

OTHER OUTCOMES:
Exploratory Objectives | Within 2 Years
  Pharmacokinetic tests to determine THIO concentration
Exploratory Objectives | Within 2 Years
  Pharmacodynamics parameters based on PCR-Based quantitative Telomeric Repeat Amplification Protocol assay in circulating tumor cells.
Exploratory Objectives | Within 2 Years
  To assess blood levels of interleukin 6.
Exploratory Objectives | Within 2 Years
  To assess blood levels of high sensitivity C-reactive protein.
Exploratory Objectives | Within 2 Years
  To assess blood levels of carcinoembryonic antigen.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Zaporojan, Medical Doctor, Study Director — MAIA Biotechnology Senior Medical Director
Locations (15):
- Centrum Medyczne Pratia, Poznan, Poland
- Romania (2):
  - Oncolab S.R.L., Craiova
  - Spitalul Clinic Municipal de Urgenta Timisoara/ Clinica de Oncologie Medicala, Timișoara
- Taiwan (8):
  - Changhua Christian Hospital (CCH), Changhua
  - Taipei Tzu Chi Hospital, Chiayi City
  - Chang-Gung Memorial Hospital - KaoHsiung, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - Chung Shan Medical University Hospital (CSMUH), Taichung
  - Taipei Medical University Hospital (TMUH), Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Gung Memorial Hospital - Linko, Taoyuan
- Turkey (Türkiye) (4):
  - Medicalpark Hastanesi, Adana
  - Liv Hospital, Ankara
  - Göztepe Süleyman Yalçın Şehir Hastanesi, Istanbul
  - İstinye University, Istanbul

IPD SHARING:
Plan to Share IPD: No